CLINICAL TRIAL: NCT00075543
Title: Phase I-II Study Of Docetaxel And Oxaliplatine In Patients With Stage III-IV Ovarian Epithelial Cancer
Brief Title: Docetaxel and Oxaliplatin in Treating Patients With Stage III or Stage IV Ovarian Epithelial Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000346887; FRE-GERCOR-DOCELOX/O-01-1; EU-20332
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-07

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel; Oxaliplatin

INTERVENTIONS:
Drug: docetaxel
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of docetaxel and oxaliplatin and to see how well they work in treating patients with stage III or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of docetaxel and oxaliplatin in patients with stage III or IV ovarian epithelial cancer.
* Determine the toxicity of this regimen in these patients.

Secondary

* Determine the tolerance profile of patients treated with this regimen.
* Determine a recommended phase III dose of this regimen in these patients.
* Determine the efficacy of this regimen, in terms of objective response rate and radiological and biological response rate (CA 125), in these patients.
* Determine the complete pathological response in patients treated with this regimen as first-line therapy.
* Determine the duration of the objective response in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive docetaxel IV over 1 hour and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 3 months.

PROJECTED ACCRUAL: A total of 30-39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial cancer

  * Stage III or IV disease
  * Metastatic peritoneal, lymphatic, or visceral disease
* Measurable or evaluable disease
* Previously untreated disease OR relapsed disease more than 6 months after the completion of a platinum-containing chemotherapy regimen
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* WHO 0-2 (0 in patients 70 to 75 years of age)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN
* Alkaline phosphatase less than 2.5 times ULN

Renal

* Creatinine no greater than 1.4 mg/dL

Other

* No serious uncontrolled infection
* No intolerance to polysorbate 80
* No peripheral neuropathy greater than grade 1
* No neurological or mental disease that would preclude study participation
* No other prior malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy
* No more than 1 prior chemotherapy regimen
* No prior oxaliplatin or docetaxel

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 28 days since prior participation in another clinical study
* No other concurrent anticancer treatment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07

PRIMARY OUTCOMES:
Maximum tolerated dose of docetaxel and oxaliplatin
Toxicity

SECONDARY OUTCOMES:
Tolerance profile
Recommended phase III dose
Efficacy
Complete pathological response
Duration of the objective response
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Tournigand, Study Chair — Hopital Saint Antoine
Locations (5):
- France (5):
  - Intercommunal Hospital, Montfermeil
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis